CLINICAL TRIAL: NCT01016457
Title: Real-Time Continuous Glucose Monitoring in Pre-School Children With Type-1 Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Kineret Mazor-Aronovitch, Ped Endocrine & Diabetes Unit, Safra's Children Hospital, Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-07-4980-KMA-CTIL
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Guardian RT — The sensor is inserted similarly to the insulin pump. It measures sub cutaneous glucose every 5 minutes. It alerts of high and low glucose levels, according to set limits.
  Other Names: Real-time continuous glucose monitoring

SUMMARY:
The purpose of this study is to compare glucose control, quality of life and number of hypoglycemias in preschool children before and after using a real-time glucosensor. Nocturnal hypoglycemia can be missed even when the parents check their children's blood glucose several times at night. The investigators hypothesise that nocturnal hypoglycemia can be prevented by using the sensor in this age group. As a consequence, quality of life of the families will improve. The investigators also hypothesise that diabetes control will improve at 3-6 months from the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Duration of diabetes for more than 6 months
* Use of insulin pump for more than 3 months

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
HbA1C | Start of study, after 3 months, after 6 months

SECONDARY OUTCOMES:
Quality of life | Before and after connecting to sensor
Number of night hypoglycemias | During 2 weeks before connecting to sensor, during connection and 3 montjs after disconnecting
Mean glucose level | During the first week of connecting to sensor and during the last week of connecting

CONTACTS AND LOCATIONS:
Overall Officials: Kineret Mazor-Aronovitch, MD, Principal Investigator
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel